CLINICAL TRIAL: NCT07249983
Title: Evaluation of SaCoVLM™ Video Laryngeal Mask Airway for Airway Management by Inexperienced Military Medics: A Two-Phase Feasibility Study
Brief Title: Evaluation of SaCoVLM™ Video Laryngeal Mask for Airway Management in Military Medics
Acronym: SAVER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Military University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Michal Soták, Principal Investigator, Charles University, Czech Republic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAVER-2025
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Airway Management; Tracheal Intubation; Anesthesia
Keywords: SaCoVLM™; Video Laryngeal Mask; Military Medic Training; Emergency Airway

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simulation and Clinical Phase (Experimental): Simulation-based and clinical use of SaCoVLM™ for airway management and intubation.
  Interventions: Device: SaCoVLM™ Video Laryngeal Mask

INTERVENTIONS:
Device: SaCoVLM™ Video Laryngeal Mask — Simulation-based and clinical use of SaCoVLM™ for airway management and intubation.

SUMMARY:
A prospective, two-phase interventional study evaluating the performance, safety, and usability of the SaCoVLM™ video laryngeal mask airway for airway management by military medics with limited intubation experience. The study includes simulation-based training and clinical application in sedated patients undergoing elective surgery.

DETAILED DESCRIPTION:
This prospective, two-phase study evaluates the use of the SaCoVLM™ video laryngeal mask airway by military medics with limited airway experience. Phase 1 involves simulated intubation on manikins to assess device placement, visualization quality, and intubation success. Phase 2 evaluates clinical performance in adult patients undergoing elective surgery under general anesthesia. Key outcomes include first-attempt success rates, insertion and intubation times, glottic visualization scores, and complication rates. The study aims to determine whether SaCoVLM™ can enable safe and effective airway management in resource-limited and prehospital military settings.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* ASA I-II
* need for airway management

Exclusion Criteria:

* Pregnancy
* known airway abnormalities
* allergy to anesthetics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
First-Attempt Success Rate of SaCoVLM™ Insertion | Within 10 minutes of airway intervention.
  Proportion of cases in which the SaCoVLM™ is successfully inserted on the first attempt during both simulated and clinical phases.
First-Attempt Success Rate of Orotracheal Intubation via SaCoVLM™ | Within 10 minutes following SaCoVLM™ placement.
  Proportion of successful orotracheal intubations on the first attempt using the SaCoVLM™ device as a conduit.

SECONDARY OUTCOMES:
Time to SaCoVLM™ Insertion | During initial airway management (simulation or clinical setting).
  Time in seconds from picking up the device to successful confirmation of placement.
Time to Successful Intubation | During initial airway management (simulation or clinical setting).
  Time in seconds from introduction of the endotracheal tube into the SaCoVLM™ to confirmed tracheal placement.
Glottic Visualization Score | Immediately after SaCoVLM™ placement.
  Laryngeal view quality assessed using Keller-Brimacombe scale. The Keller-Brimacombe score ranges from Grade 1 (vocal cords not visible) to Grade 4 (only vocal cords visible with a full, unobstructed view), with higher grades indicating better glottic visualization and alignment for intubation.
Subjective Difficulty Score | Immediately after each procedure.
  Operator-rated difficulty of device use on a 10-point visual analog scale (VAS).
Incidence of Airway Complications | From initiation of airway management to induction of general anesthesia (clinical phase only).
  Number of adverse airway events including hypoxemia (SpO₂ < 90%), laryngospasm, or aspiration.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Sotak, M.D., Ph.D., Principal Investigator — Military University Hospital, Prague
Locations (1):
- Military University Hospital Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mishra N, Bharadwaj A. Comparison of Fiberoptic-Guided Tracheal Intubation Through Intubating Laryngeal Mask Airway (ILMA) FastrachTM and Ambu(R) Aura-i: A Randomized Clinical Study. Cureus. 2020 Sep 1;12(9):e10178. doi: 10.7759/cureus.10178. PMID 33029458